CLINICAL TRIAL: NCT02394184
Title: Evaluation of Clinical Outcomes of Transcatheter Aortic Valve Replacement for Patients With Bicuspid Aortic Valve Stenosis
Brief Title: The Bicuspid Aortic Stenosis Following Transcatheter Aortic Valve Replacement Registry
Acronym: Bicuspid TAVR
Status: Completed | Type: Observational
Sponsor: Seung-Jung Park (Other)
Collaborators: CardioVascular Research Foundation, Korea (Other)
Responsible Party: Sponsor-Investigator, Seung-Jung Park, MD, PhD, Asan Medical Center
Organization: Asan Medical Center (Other)
Other Study IDs: AMCCV2014-14_sub
Record Dates: First submitted 2015-03-09; First posted 2015-03-20 (Estimated); Last update posted 2019-12-26 (Actual); Status verified 2019-12

CONDITIONS: Aortic Valve Stenosis; Cardiovascular Diseases; Heart Valve Diseases; Bicuspid
Keywords: transcatheter aortic valve replacement
MeSH Terms: conditions — Aortic Valve Stenosis; Cardiovascular Diseases; Heart Valve Diseases; Bicuspid Aortic Valve Disease | interventions — Transcatheter Aortic Valve Replacement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- patients with bicuspid aortic valve stenosis
  Interventions: Procedure: transcatheter aortic valve replacement

INTERVENTIONS:
Procedure: transcatheter aortic valve replacement

SUMMARY:
The purpose of this study is to evaluate the clinical outcomes of transcatheter aortic valve replacement (TAVR) in patients with bicuspid aortic valve stenosis.

DETAILED DESCRIPTION:
This registry is a subgroup of Asian TAVR registry(NCT02308150) and Asian TAVR registry changes to TP-TAVR registry(NCT03826264). Some subjects moved to TP-TAVR registry and continue to 10-year follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Patients with bicuspid aortic valve stenosis who are not candidates for surgical aortic valve replacement because of coexisting illnesses.
* The patient or guardian agrees to the study protocol and the schedule of clinical follow-up, and provides informed, written consent, as approved by the appropriate Institutional Review Board/Ethics Committee of the respective clinical site.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients with bicuspid aortic valve stenosis
Sampling Method: Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2015-05; Primary Completion 2019-09-24 (Actual); Study Completion 2019-09-24 (Actual)

PRIMARY OUTCOMES:
Death | 1 month
Death | 6 months
Death | 1 year
Death | 2 years
Death | 3 years
Death | 4 years
Death | 5 years

SECONDARY OUTCOMES:
Death from cardiac cause | 1 month
Death from cardiac cause | 6 months
Death from cardiac cause | 1 year
Death from cardiac cause | 2 years
Death from cardiac cause | 3 years
Death from cardiac cause | 4 years
Death from cardiac cause | 5 years
Stroke | 1 month
Stroke | 6 months
Stroke | 1 year
Stroke | 2 years
Stroke | 3 years
Stroke | 4 years
Stroke | 5 years
Myocardial infarction | 1 month
Myocardial infarction | 6 months
Myocardial infarction | 1 year
Myocardial infarction | 2 years
Myocardial infarction | 3 years
Myocardial infarction | 4 years
Myocardial infarction | 5 years
Repeat hospitalization | 1 month
Repeat hospitalization | 6 months
Repeat hospitalization | 1 year
Repeat hospitalization | 2 years
Repeat hospitalization | 3 years
Repeat hospitalization | 4 years
Repeat hospitalization | 5 years
Acute kidney injury | 1 month
Acute kidney injury | 6 months
Acute kidney injury | 1 year
Acute kidney injury | 2 years
Acute kidney injury | 3 years
Acute kidney injury | 4 years
Acute kidney injury | 5 years
Vascular complication | 1 month
Vascular complication | 6 months
Vascular complication | 1 year
Vascular complication | 2 years
Vascular complication | 3 years
Vascular complication | 4 years
Vascular complication | 5 years
Bleeding events | 1 month
Bleeding events | 6 months
Bleeding events | 1 year
Bleeding events | 2 years
Bleeding events | 3 years
Bleeding events | 4 years
Bleeding events | 5 years
Device success | 1 month
Device success | 6 months
Device success | 1 year
Device success | 2 years
Device success | 3 years
Device success | 4 years
Device success | 5 years
Early safety as a composite of all cause mortality, all stroke, life threatening bleeding, acute kidney injury, coronary artery obstruction requiring intervention, major vascular complication, valve related dysfunction requiring repeat procedure | 1 month
Clinical Efficacy as a composite of all cause mortality, all stroke, hospitalization for valve related symptoms or worsening congestive heart failure, NYHA class III or IV, prosthetic heart valve dysfunction | 1 month, 6 months, and annually at 1 to 5 years
Time related valve safety as a composite of structural valve deterioration, prosthetic valve endocarditis, prosthetic valve thrombosis, thromboembolic events, VARC bleeding(unless clearly unrelated to valve therapy) | from index procedure to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Seung-jung Park, MD, PhD, Principal Investigator — Division of Cardiology, Department of Medicine, Heart Institute, Asan Medical Center, University of Ulsan College of Medicine; Gerald Yong, MD, Principal Investigator — Perth Cardiovascular Institute, Royal Perth Hospital 197 Wellington Street, Perth WA 6000, Australia; Edgar Tay, MD, Principal Investigator — Department of Cardiology, National University Hospital Singapore, 5 Lower Kent Ridge Road, Singapore 119074, Singapore; Fabian Nietlispach, MD, PhD, Principal Investigator — Department of Cardiology, University Heart Center, Raemistrasse 100, CH-8091 Zurich, Switzerland; Corrado Tamburino, MD, Principal Investigator — Division of Cardiology, Ferrarotto Hospital, University of Catania; ETNA Foundation Via Citelli 6, 95124, Catania, Italy; Thierry Lefèvre, MD, Principal Investigator — Institut Hospitalier Jacques Cartier, 6 avenue du Noyer Lambert, FR-91300 Massy, France; Marie-Claude Morice, MD, Principal Investigator — Institut Hospitalier Jacques Cartier, 6 avenue du Noyer Lambert, FR-91300 Massy, France; Jeroen J. Bax, MD, PhD, Principal Investigator — Department of Cardiology, Leiden University Medical Center, Albinusdreef 2, 2300 RC, Leiden, The Netherlands; John G. Webb, MD, Principal Investigator — St. Paul's Hospital, University of British Columbia, 1081 Burrard Street, Vancouver, BC V6Z 1Y6, Canada; Susheel Kodali, MD, Principal Investigator — Herbert and Sandi Feinberg Interventional Cardiology, Heart Valve Center at Columbia University Medical Center/New York-Presbyterian Hospital, 177 Fort Washington Avenue,
Locations (1):
- Asan Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No
This is not a publicly funded trial.

REFERENCES:
- [Derived] Yoon SH, Lefevre T, Ahn JM, Perlman GY, Dvir D, Latib A, Barbanti M, Deuschl F, De Backer O, Blanke P, Modine T, Pache G, Neumann FJ, Ruile P, Arai T, Ohno Y, Kaneko H, Tay E, Schofer N, Holy EW, Luk NHV, Yong G, Lu Q, Kong WKF, Hon J, Kao HL, Lee M, Yin WH, Park DW, Kang SJ, Lee SW, Kim YH, Lee CW, Park SW, Kim HS, Butter C, Khalique OK, Schaefer U, Nietlispach F, Kodali SK, Leon MB, Ye J, Chevalier B, Leipsic J, Delgado V, Bax JJ, Tamburino C, Colombo A, Sondergaard L, Webb JG, Park SJ. Transcatheter Aortic Valve Replacement With Early- and New-Generation Devices in Bicuspid Aortic Valve Stenosis. J Am Coll Cardiol. 2016 Sep 13;68(11):1195-1205. doi: 10.1016/j.jacc.2016.06.041. PMID 27609682